CLINICAL TRIAL: NCT01432743
Title: Cartomerge Versus NavX Fusion in Catheter Ablation of Atrial Fibrillation
Acronym: CAVERN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Principal Investigator, Dr Richard Schilling, Professor of Cardiology and Cardiac Electrophysiology, Barts & The London NHS Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 005126
Record Dates: First submitted 2011-02-21; First posted 2011-09-13 (Estimated); Last update posted 2011-09-13 (Estimated); Status verified 2011-09

CONDITIONS: Atrial Fibrillation
Keywords: 3D mapping; Image integration; Atrial fibrillation; Catheter Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cartomerge (Experimental): Use of Cartomerge to guide ablation
  Interventions: Procedure: Cartomerge
- NavX Fusion (Active Comparator): Use of NavX fusion to guide ablation
  Interventions: Procedure: NavX Fusion

INTERVENTIONS:
Procedure: NavX Fusion — Using NavX Fusion to guide catheter ablation
  Other Names: NavX Fusion (St Jude) - electroanatomic mapping
  Arms: NavX Fusion
Procedure: Cartomerge — Guidance of catheter ablation using Cartomerge guidance
  Other Names: Cartomerge (Biosense Webster) - electroanatomic mapping
  Arms: Cartomerge

SUMMARY:
Comparison of Two Strategies for Catheter Ablation of Atrial Fibrillation - a comparison of ablation guided by Cartomerge and NavX Fusion. 3D mapping systems are widely used in catheter ablation of AF. Integration of a previously acquired image of the left atrium into the electroanatomical (EA) map offers several potential advantages, including visualisation of the complex anatomy of the left atrium, reduction of fluoroscopy time and improved results . The two most widely used systems are Cartomerge (Biosense Webster, etc) and NavX Fusion (SJM, etc). Although both systems have been independently validated, their clinical utility has not previously been directly compared in a randomised trial

DETAILED DESCRIPTION:
Patients are randomised to either NavX Fusion or Cartomerge. They undergo a standard catheter ablation procedure and data is collected. Both systems are routinely used in our clinical practise. This is a comparison trial of 2 mapping technologies.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age
* Be undergoing their first planned procedure for electrophysiology mapping and ablation in the left atrium of AF
* Be willing and able to sign the study specific informed consent
* Have a negative pregnancy test for female subjects of child bearing potential

Exclusion Criteria:

* Have a left ventricular ejection fraction (LVEF) of <40% as evaluated by pre-procedure TTE
* Have any contraindication or allergy to routine procedural medications or catheter materials
* Have any condition for which the investigator feels it is unsafe for the subject to undergo an invasive electrophysiology procedure (EP) catheterisation
* Be currently participating in another clinical research study
* Have any condition for which the subject's life expectancy is less than twelve months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2007-09; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
AF recurrence | 6 months
  Documentation of symptomatic arrhythmia or arrhythmia on a 7 day holter monitor at six-month follow-up

SECONDARY OUTCOMES:
Lesion distance from CT shell | At completion of catheter ablation procedure (distance at defined procedure endpoint) (between 0 - 6 hours after procedure start)
  Establish accuracy of lesion placement in relation to previously acquired CT shell to act as an indicator of guidance accuracy
Procedural time points | At start, during and end of inpatient catheter ablation procedure. (between 0 & 6 hours after start of ablation procedure)
  Measurement of all procedural time points during procedure, along with x-ray dose and screening times.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Schilling, FRCP, Principal Investigator — Barts and the London NHS Trust
Locations (1):
- Barts and the London NHS Trust, London, United Kingdom

REFERENCES:
- [Derived] Finlay MC, Hunter RJ, Baker V, Richmond L, Goromonzi F, Thomas G, Rajappan K, Duncan E, Tayebjee M, Dhinoja M, Sporton S, Earley MJ, Schilling RJ. A randomised comparison of Cartomerge vs. NavX fusion in the catheter ablation of atrial fibrillation: the CAVERN Trial. J Interv Card Electrophysiol. 2012 Mar;33(2):161-9. doi: 10.1007/s10840-011-9632-7. Epub 2011 Nov 26. PMID 22119854